CLINICAL TRIAL: NCT06907329
Title: The Impact of Nicotinamide Mononucleotide Sustained-release Tablets on Immunosenescence and Metablism in Middle-aged and Elderly Individuals With Metabolic Disorders.
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Qing Su (Other)
Responsible Party: Sponsor-Investigator, Qing Su, Director, Dept of Endocrinology,Xinhua Hospital, Xinhua Hospital, Shanghai Jiao Tong University School of Medicine
Organization: Xinhua Hospital, Shanghai Jiao Tong University School of Medicine (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: XHEC-C-2024-165-4
Record Dates: First submitted 2025-03-19; First posted 2025-04-02 (Actual); Last update posted 2025-07-08 (Actual); Status verified 2025-06

CONDITIONS: Immunosenescence; Metabolism

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- NMN Arm (Experimental): NMN tablets (1000mg/tablet) , 1 tablet daily before breakfast
  Interventions: Dietary Supplement: NMN
- Placebo Arm (Placebo Comparator): Matching Placebo (tablets) once daily before breakfast
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: NMN — NMN SR tablets(1000mg/tablets) , 1 tablet daily before breakfast
  Arms: NMN Arm
Dietary Supplement: Placebo — Matching Placebo (tablets) once daily before breakfast
  Arms: Placebo Arm

SUMMARY:
The ageing of our country is increasing and the ageing of the population has led to a significant increase in aging related diseases. During the aging process of the organism, cellular senescence can occur in all systems of the body, of which the senescence of the immune system is called immunosenescence. Some studies have shown that metabolic disorders can also trigger aging. This study investigated the effect of nicotinamide mononucleotide (NMN) supplementation on immunosenescence in middle-aged and elderly people through a placebo-controlled long-range clinical trail, aiming to provide a new method to improve immunosenescence. The effects of NMN supplementation on glucose and lipid metabolic indexes, body composition and telomere length of peripheral blood cells are also investigated, which may open up new ideas for the prevention and treatment of glucose and lipid metabolic diseases.

DETAILED DESCRIPTION:
A randomised, placebo-controlled, parallel group study to assess the efficacy and safety of NMN in middle-aged and elderly people with immunosenescence. People aged 50-70 years will be included in the study. Participants will be given NMN SR tablets (1000mg/tablet) or placebo, 1 tablet daily before breakfast. The study treatment period lasts 26 weeks. Investigator visits will be conducted at months 1, 3 and 6. Percentage of CD3+CD8+CD27-CD28- cells to total CD3+CD8+ T cells will be used as the primary evaluation metrics for assessing efficacy.Liver fat content, body composition analysis, pancreatic β-cell function, telomere length, fasting blood glucose, glycosylated hemoglobin, and cardiorespiratory fitness will be used as secondary indicators for efficacy assessment. Physiological and biochemical parameters such as blood and urine routine, liver and kidney function will be used for safety assessment.

ELIGIBILITY:
Inclusion Criteria:

1. Age 50-70 years with overweight or obesity (BMI 24kg/m2);
2. At least one of the following three: metabolism-related fatty liver disease (diagnosed by ultrasound); pre-diabetes; type 2 diabetes mellitus with HbA1c <7% without glucose-lowering drug therapy;
3. Agreed to participate in the trial and could adhere to the follow-up and visit the hospital on their own; signed the informed consent form.

Exclusion Criteria:

1. Patients with tumours;
2. Patients with autoimmune diseases (excluding Hashimoto's thyroiditis);
3. Severe cardiovascular disease or cardiac insufficiency;
4. Systolic blood pressure > 160 mmHg or diastolic blood pressure > 100 mmHg;
5. Chronic obstructive pulmonary disease;
6. Chronic active hepatitis or cirrhosis;
7. Chronic renal insufficiency;
8. Stroke patients
9. Severe haematological diseases;
10. Infectious diseases;
11. Mental illness;
12. Other conditions that, in the opinion of the investigator, may affect the results of the study;
13. Those who have used NMN or other anti-aging agents within six months.
14. Premenopausal woman
15. ALT, AST values are more than three times higher than the upper limit of the normal reference range

Ages: 50 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 126 (Estimated)
Dates: Start 2025-06-05 (Actual); Primary Completion 2027-03-31 (Estimated); Study Completion 2027-03-31 (Estimated)

PRIMARY OUTCOMES:
CD3+CD8+CD27-CD28- T cells as a percentage of CD3+CD8+ T cells, expressed in %, evaluated by flow cytometry | 26 weeks

SECONDARY OUTCOMES:
Body composition analysis, expressed in kg, %, and g/cm², evaluated by dual-energy X-ray absorptiometry | 26 weeks
Determination of fasting blood glucose and OGTT 2-hour blood glucose, expressed in mmol/L, evaluated by glucose oxidase method | 26 weeks
CD3+CD8+CD27- T cells as a percentage of total CD3+CD8+ T cells, expressed in %, evaluated by flow cytometry | 26 weeks
CD3+CD8+CD28- T cells as a percentage of total CD3+CD8+ T cells, expressed in %, evaluated by flow cytometry | 26 weeks
CD3+CD4+CD27- T cells as a percentage of CD3+CD4+ T cells, expressed in %, evaluated by flow cytometry | 26 weeks
CD3+CD4+CD28- T cells as a percentage of CD3+CD4+ T cells, expressed in %, evaluated by flow cytometry | 26 weeks
CD3+CD4+CD27-CD28- T cells as a percentage of CD3+CD4+ T cells, expressed in %, evaluated by flow cytometry | 26 weeks
CD3+CD8+CD45RA+CCR7- T cells as a percentage of CD3+CD8+ T cells, expressed in %, evaluated by flow cytometry | 26 weeks
CD3+CD8+CD57+KLRG1+ T cells as a percentage of CD3+CD8+ T cells, expressed in %, evaluated by flow cytometry | 26 weeks
CD3+CD8+ T cells as a percentage of CD3+CD4+ T cells, expressed in %, evaluated by flow cytometry | 26 weeks
NMN, NAD+ levels in peripheral blood cells, evaluated by mass spectrometry | 26 weeks
Peripheral blood cell telomere length, expressed as a unitless value , evaluated by Quantitative Real-time polymerase chain reaction | 26 weeks
Cardiorespiratory fitness related indicators, expressed in mL/kg/min, L/min, beats/min, and unitless ratios, evaluated by COSMED metabolic cart during cardiopulmonary exercise testing | 26 weeks
Glycosylated hemoglobin, expressed in mmol/mol, evaluated by HPLC | 26 weeks
Pancreatic β-cell function, expressed as a unitless value, evaluated by HOMA-β、HOMA-IR | 26 weeks
Weight, expressed in kilograms, evaluated by weighing scale | 26 weeks
Waist circumference, expressed in centimeters, evaluated by tape measure | 26 weeks
Waist-to-hip ratio, expressed as a unitless ratio, evaluated using a standardized tape measure following WHO measurement protocols. | 26 weeks
Waist-to-height, expressed as a unitless ratio, evaluated using a standardized tape measure following WHO measurement protocols. | 26 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Xin Hua Hospital Affiliated to Shanghai Jiao Tong University School of Medicine, Shanghai, China

IPD SHARING:
Plan to Share IPD: No